CLINICAL TRIAL: NCT00117325
Title: A 4 Week Randomized, Double Blind, Placebo Controlled Study of GW685698X Aq Nasal Spray 100mcg QD in Adults and Adolescents With Vasomotor Rhinitis
Brief Title: Study Of Adults And Adolescents With Vasomotor Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: FFR30006
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Vasomotor
Keywords: Vasomotor Rhinitis; VMR; nonallergic rhinitis; GW685698X
MeSH Terms: conditions — Rhinitis, Vasomotor

ARMS (1):
- GW685698X (Experimental): GW685698X
  Interventions: Drug: GW685698X

INTERVENTIONS:
Drug: GW685698X — Aqueous Nasal Spray 100mcg

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of GW685698X 100mcg once daily (QD) aqueous nasal spray with vehicle placebo nasal spray in adult and adolescent subjects (12 years of age and older) with vasomotor rhinitis (VMR).

ELIGIBILITY:
Inclusion criteria:

* Must be outpatients.
* Diagnosis of VMR.
* Literate in English or native language.

Exclusion criteria:

* Significant concomitant medical condition.
* Use corticosteroids or other allergy medications during the study.
* Used tobacco products within the past year.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2005-07-11 (Actual); Primary Completion 2006-02-09 (Actual); Study Completion 2006-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (37):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Barbara, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Ypsilanti, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Mount Laurel, New Jersey
  - GSK Investigational Site, Liverpool, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, North Olmsted, Ohio
  - GSK Investigational Site, Lake Oswego, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Easton, Pennsylvania
  - GSK Investigational Site, Palmyra, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Salt Lake City, Utah
- Canada (3):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Québec
- Czechia (3):
  - GSK Investigational Site, Litoměřice
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Tábor
- Germany (5):
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Hamburg
- Norway (2):
  - GSK Investigational Site, Larvik
  - GSK Investigational Site, Nesttun
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Deva

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: FFR30006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The actual dose delivered from the product was 27.5 micrograms (µg) /actuation, which is therefore proposed as the label claim rather than 25 µg/actuation. Based on this spray content assessment, the dose examined in this study was actually 110 µg rather than the 100 µg dose indicated in the protocol.
Pre-assignment Details: Out of 901 participants screened, 549 participants were screen failures and hence were not randomized into the study. Out of 901 participants screened, 352 participants were randomized from 11 July 2005 to 16 January 2006.
Groups:
- Placebo: Participants received placebo matching with GW685698X aqueous nasal spray 110 microgram (mcg) administered as two sprays from the device into each nostril once daily every morning up to 4 weeks.
- Fluticasone Furoate 110 mcg QD: Participants received Fluticasone Furoate (GW 685698X) aqueous nasal spray 110 mcg administered as two sprays from the device into each nostril once daily every morning up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Started | 173 | 179
Completed | 160 | 167
Not Completed | 13 | 12
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Use of prohibited medicine | 1 | 2
Not completed — Early termination | 1 | 1
Not completed — Admisnitrative | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received placebo matching with GW685698X aqueous nasal spray 110 mcg administered as two sprays from the device into each nostril once daily every morning up to 4 weeks.
- Fluticasone Furoate 110 mcg QD: Participants received GW685698X aqueous nasal spray 110 mcg administered as two sprays from the device into each nostril once daily every morning up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD | Total
Number analyzed (Participants) | 173 | 179 | 352
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (14.66) | 46.6 (16.77) | 45.8 (15.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 125 | 247
  Male | 51 | 54 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 163 | 169 | 332
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Daily Reflective Total Nasal Symptom Score (rTNSS)
Description: The daily rTNSS was the average of the AM (morning) and PM (before bed time) rTNSS assessments. Each rTNSS assessment comprised the sum of the three nasal symptom scores for rhinorrhea, nasal congestion and postnasal drip where each symptom was scored on a scale of 0 (no symptoms) to 3 (severe symptoms).. The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: Due to irregularities found during a compliance audit, a reduced intent-to-treat (RITT) population was defined which excludes two participants from one of the investigative sites.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 170 | 176
Score on scale | -1.71 (0.16) | -2.05 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD Week 1-4 analysis; Test type: Superiority or Other; p = 0.050, ANCOVA; Analysis of covariance (ANCOVA) method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.335, 95% CI 2-sided [-0.67 to 0.00]

2. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Morning (AM), Pre-dose, Instantaneous Total Nasal Symptom Scores (iTNSS)
Description: The AM, pre-dose, iTNSS is the sum of the 3 individual nasal symptom score assessments for rhinorrhea, nasal congestion and postnasal drip performed at the moment immediately prior to taking their dose where each symptom was scored on a scale of 0 to 3 (0= no symptoms, 3= severe symptoms). . The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. Change from baseline was calculated as endpoint value minus the baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: Reduced ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 170 | 176
Score on scale | -1.48 (0.16) | -1.87 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD Week 1-4 analysis; Test type: Superiority or Other; p = 0.027, ANCOVA — Week 1-4; ANCOVA method was used adjusting for baseline iTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.393, 95% CI 2-sided [-0.74 to -0.05]

3. Secondary Outcome: Number of Participants With Overall Evaluation of Response to Therapy
Description: The overall evaluation of Response to Therapy was based on a 7-point categorical scale where the participants rated their perception of the change or lack of change in their VMR (Vasomotor rhinitis) symptoms at the end of the study. The 7 categories were: 1=significantly improved, 2=moderately improved, 3= mildly improved, 4= no change, 5= mildly worse, 6= moderately worse, and 7= significantly worse.
Time Frame: Up to 4 weeks
Population: RITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 168 | 176
Participants
  Significantly Improved | 26 | 33
  Moderately Improved | 37 | 40
  Mildly Improved | 45 | 47
  No Change | 52 | 50
  Mildly Worse | 1 | 3
  Moderately Worse | 4 | 1
  Significantly Worse | 3 | 2
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD up to Week 4 analysis; Test type: Superiority or Other; p = 0.184, Regression, Logistic; logistic regression adjusting for age, gender, investigator, and treatment; Effectiveness of study medication for relieving non-allergic rhinitis symptoms over the entire treatment period (Total response) was analyzed

4. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in AM Pre-dose rTNSS
Description: The rTNSS is a rating of the severity of symptoms over the previous 12 hours and is performed in the AM (AM rTNSS). . The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. The TNSS was the sum of the individual symptom scores for rhinorrhoea, nasal congestion and post-nasal drip which was scored on a scale of 0-3. Change from Baseline was calculated as post randomization value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 170 | 176
Score on scale | -1.69 (0.16) | -2.04 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD Week 1-4 analysis; Test type: Superiority or Other; p = 0.051, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.348, 95% CI 2-sided [-0.70 to 0.00]

5. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Evening (PM) rTNSS
Description: The TNSS was the sum of the individual symptom scores for rhinorrhoea, nasal congestion and post-nasal drip which was scored on a scale of 0-3. The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. The rTNSS is a rating of the severity of symptoms over the previous 12 hours and is performed in the PM (PM rTNSS). Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale | -1.77 (0.16) | -2.07 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD up to Week 4 analysis; Test type: Superiority or Other; p = 0.076, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.304, 95% CI 2-sided [-0.64 to 0.03]

6. Secondary Outcome: Mean Percent Change From Baseline Over the Entire Treatment Period in Daily rTNSS
Description: The daily rTNSS was the average of the AM (morning) and PM (before bed time) rTNSS assessments.The TNSS was the sum of the individual symptom scores for rhinorrhoea, nasal congestion and post-nasal drip which was scored on a scale of 0-3. The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change in score
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 170 | 176
Percent change in score | -26.14 (2.45) | -30.65 (2.40)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD Week 1-4 analysis; Test type: Superiority or Other; p = 0.093, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -4.510, 95% CI 2-sided [-9.77 to 0.75]

7. Secondary Outcome: Mean Percent Change From Baseline Over the Entire Treatment Period in AM, Pre-dose iTNSS
Description: The AM, pre-dose, iTNSS is the sum of the 3 individual nasal symptom score assessments for rhinorrhea, nasal congestion and postnasal drip performed at the moment immediately prior to taking their dose where each symptom was scored on a scale of 0 to 3. The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change in score
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 170 | 176
Percent change in score | -21.09 (2.54) | -27.46 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD Week 1-4 analysis; Test type: Superiority or Other; p = 0.023, ANCOVA; ANCOVA method was used adjusting for baseline iTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -6.372, 95% CI 2-sided [-11.8 to -0.90]

8. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Individual Daily, Reflective Nasal Symptom Scores for Rhinorrhea, Nasal Congestion and Post-nasal Drip
Description: The TNSS was the sum of the individual symptom scores for rhinorrhoea, nasal congestion and post-nasal drip which was scored on a scale of 0-3. The severity of symptoms was defined as 0: none-symptom was not present, 1: mild-sign/symptom was clearly present but minimal awareness; easily tolerated, 2: moderate-definite awareness of sign/symptom that was bothersome but tolerable, 3: severe (sign/symptom was hard to tolerate; causes interference with activities of daily living and/or sleeping. The daily reflective nasal symptom scores was the average of the AM (morning) and PM (before bed time) rTNSS assessments. Each rTNSS assessment comprised the sum of the three nasal symptom. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale
  Rhinorrhea: number analyzed (Participants) | 170 | 176
  Rhinorrhea | -0.50 (0.06) | -0.62 (0.06)
  Nasal Congestion: number analyzed (Participants) | 170 | 176
  Nasal Congestion | -0.68 (0.06) | -0.81 (0.06)
  Post-nasal Drip: number analyzed (Participants) | 171 | 176
  Post-nasal Drip | -0.51 (0.06) | -0.61 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for Rhinorrhea; Test type: Superiority or Other; p = 0.061, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.118, 95% CI 2-sided [-0.24 to 0.01]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for Nasal Congestion; Test type: Superiority or Other; p = 0.061, ANCOVA; Mean Difference (Net) = -0.124, 95% CI 2-sided [-0.25 to 0.01]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for post-nasal drip; Test type: Superiority or Other; p = 0.138, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.095, 95% CI 2-sided [-0.22 to 0.03]

9. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Individual AM, Pre-dose, Instantaneous, Nasal Symptom Scores for Rhinorrhea, Nasal Congestion and Postnasal Drip
Description: The AM, pre-dose, instantaneous nasal symptom score is the sum of the 3 individual nasal symptom score assessments for rhinorrhea, nasal congestion and postnasal drip performed at the moment immediately prior to taking their dose where each symptom was scored on a scale of 0 to 3 (0= no symptoms, 3= severe symptoms). Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale
  Rhinorrhea: number analyzed (Participants) | 170 | 176
  Rhinorrhea | -0.44 (0.06) | -0.56 (0.06)
  Nasal congestion: number analyzed (Participants) | 170 | 176
  Nasal congestion | -0.54 (0.06) | -0.70 (0.06)
  Post-nasal drip: number analyzed (Participants) | 170 | 176
  Post-nasal drip | -0.48 (0.06) | -0.60 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for Rhinorrhea; Test type: Superiority or Other; p = 0.087, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.113, 95% CI 2-sided [-0.24 to 0.02]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for nasal congestion; Test type: Superiority or Other; p = 0.015, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.164, 95% CI 2-sided [-0.30 to -0.03]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for post-nasal drip; Test type: Superiority or Other; p = 0.106, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.112, 95% CI 2-sided [-0.25 to 0.02]

10. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Individual AM, Reflective Nasal Symptom Scores for Rhinorrhea, Nasal Congestion and Postnasal Drip
Description: The reflective nasal symptom score is a rating of the severity of symptoms over the previous 12 hours and is performed in the AM (AM rTNSS). Score assessments for rhinorrhea, nasal congestion and postnasal drip performed at the moment immediately prior to taking their dose where each symptom was scored on a scale of 0 to 3 (0= no symptoms, 3= severe symptoms). Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Groups:
- Fluticasone Furoate 110mcg QD: Participants received GW685698X aqueous nasal spray 110 mcg administered as two sprays from the device into each nostril once daily every morning up to 4 weeks.
Arm/Group | Placebo | Fluticasone Furoate 110mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale
  Rhinorrhea: number analyzed (Participants) | 170 | 176
  Rhinorrhea | -0.48 (0.06) | -0.61 (0.06)
  Nasal congestion: number analyzed (Participants) | 170 | 176
  Nasal congestion | -0.65 (0.06) | -0.78 (0.06)
  Post-nasal drip: number analyzed (Participants) | 170 | 176
  Post-nasal drip | -0.55 (0.06) | -0.64 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rhinorrhea; Test type: Superiority or Other; p = 0.048, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.132, 95% CI 2-sided [-0.26 to -0.00]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for Nasal congestion; Test type: Superiority or Other; p = 0.076, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.124, 95% CI 2-sided [-0.26 to 0.01]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 110mcg QD; Placebo versus Fluticasone Furoate 110 mcg for post-nasal drip; Test type: Superiority or Other; p = 0.164, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.093, 95% CI 2-sided [-0.22 to 0.04]

11. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in Individual PM, Reflective, Nasal Symptom Scores for Rhinorrhea, Nasal Congestion and Postnasal Drip
Description: The reflective nasal symptom score is a rating of the severity of symptoms over the previous 12 hours and was performed in the PM (PM rTNSS). Score assessments for rhinorrhea, nasal congestion and postnasal drip performed at the moment immediately prior to taking their dose where each symptom was scored on a scale of 0 to 3 (0= no symptoms, 3= severe symptoms). Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and up to Week 4
Population: RITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale
  Rhinorrhea: number analyzed (Participants) | 170 | 176
  Rhinorrhea | -0.53 (0.06) | -0.59 (0.06)
  Nasal congestion: number analyzed (Participants) | 170 | 176
  Nasal congestion | -0.73 (0.06) | -0.84 (0.06)
  Post-nasal drip: number analyzed (Participants) | 171 | 176
  Post-nasal drip | -0.49 (0.06) | -0.59 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for Rhinorrhea; Test type: Superiority or Other; p = 0.136, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.096, 95% CI 2-sided [-0.22 to 0.03]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for nasal congestion; Test type: Superiority or Other; p = 0.100, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.111, 95% CI [-0.24 to 0.02]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for post-nasal drip; Test type: Superiority or Other; p = 0.100, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.111, 95% CI 2-sided [-0.24 to 0.02]

12. Secondary Outcome: Mean Scores Changes From Baseline as a Function of Time
Description: The onset of treatment effect was assessed by the mean change from Baseline in AM iTNSS (Days 1 to 28), the mean change from Baseline in daily rTNSS (Days 1 to 28), and mean change from Baseline in AM rTNSS and PM rTNSS. The time to maximum effect was also evaluated by the mean change from Baseline in daily rTNSS for Days 1 to 28. Change from Baseline was calculated as any post-Baseline value minus the Baseline value. Baseline visit was 4 days prior to randomization (Day 1).
Time Frame: Baseline (4 days prior to randomization [Day 1]) and Daily for 28 days
Population: RITT population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Fluticasone Furoate 110 mcg QD
Number analyzed (Participants) | 172 | 178
Score on scale
  AM iTNSS Day 1: number analyzed (Participants) | 165 | 175
  AM iTNSS Day 1 | -0.47 (0.16) | -0.92 (0.16)
  AM iTNSS Day 2: number analyzed (Participants) | 166 | 173
  AM iTNSS Day 2 | -0.69 (0.17) | -1.01 (0.17)
  AM iTNSS Day 3: number analyzed (Participants) | 167 | 175
  AM iTNSS Day 3 | -0.75 (0.18) | -1.14 (0.18)
  AM iTNSS Day 4: number analyzed (Participants) | 167 | 173
  AM iTNSS Day 4 | -0.96 (0.18) | -1.22 (0.18)
  AM iTNSS Day 5: number analyzed (Participants) | 165 | 172
  AM iTNSS Day 5 | -1.15 (0.20) | -1.45 (0.19)
  AM iTNSS Day 6: number analyzed (Participants) | 166 | 174
  AM iTNSS Day 6 | -1.01 (0.20) | -1.59 (0.19)
  AM iTNSS Day 7: number analyzed (Participants) | 166 | 175
  AM iTNSS Day 7 | -1.17 (0.20) | -1.55 (0.19)
  AM iTNSS Day 8: number analyzed (Participants) | 165 | 170
  AM iTNSS Day 8 | -1.38 (0.20) | -1.61 (0.20)
  AM iTNSS Day 9: number analyzed (Participants) | 163 | 169
  AM iTNSS Day 9 | -1.47 (0.20) | -1.66 (0.20)
  AM iTNSS Day 10: number analyzed (Participants) | 161 | 169
  AM iTNSS Day 10 | -1.31 (0.21) | -1.78 (0.21)
  AM iTNSS Day 11: number analyzed (Participants) | 160 | 169
  AM iTNSS Day 11 | -1.48 (0.22) | -1.66 (0.21)
  AMiTNSS Day 12: number analyzed (Participants) | 159 | 168
  AMiTNSS Day 12 | -1.52 (0.22) | -1.86 (0.21)
  AM iTNSS Day 13: number analyzed (Participants) | 158 | 168
  AM iTNSS Day 13 | -1.48 (0.22) | -1.83 (0.21)
  AM iTNSS Day 14: number analyzed (Participants) | 160 | 165
  AM iTNSS Day 14 | -1.72 (0.21) | -1.95 (0.20)
  AM iTNSS Day 15: number analyzed (Participants) | 163 | 163
  AM iTNSS Day 15 | -1.54 (0.21) | -1.92 (0.21)
  AM iTNSS Day 16: number analyzed (Participants) | 163 | 165
  AM iTNSS Day 16 | -1.56 (0.21) | -1.99 (0.21)
  AM iTNSS Day 17: number analyzed (Participants) | 161 | 162
  AM iTNSS Day 17 | -1.64 (0.22) | -2.20 (0.22)
  AM iTNSS Day 18: number analyzed (Participants) | 162 | 164
  AM iTNSS Day 18 | -1.75 (0.21) | -2.21 (0.21)
  AM iTNSS Day 19: number analyzed (Participants) | 162 | 165
  AM iTNSS Day 19 | -1.70 (0.21) | -2.33 (0.21)
  AM iTNSS Day 20: number analyzed (Participants) | 157 | 165
  AM iTNSS Day 20 | -1.89 (0.22) | -2.11 (0.21)
  AM iTNSS Day 21: number analyzed (Participants) | 158 | 161
  AM iTNSS Day 21 | -1.97 (0.22) | -2.26 (0.22)
  AM iTNSS Day 22: number analyzed (Participants) | 154 | 164
  AM iTNSS Day 22 | -1.73 (0.22) | -2.32 (0.22)
  AM iTNSS Day 23: number analyzed (Participants) | 157 | 164
  AM iTNSS Day 23 | -1.80 (0.23) | -2.27 (0.22)
  AM iTNSS Day 24: number analyzed (Participants) | 157 | 165
  AM iTNSS Day 24 | -1.93 (0.23) | -2.40 (0.22)
  AM iTNSS Day 25: number analyzed (Participants) | 156 | 164
  AM iTNSS Day 25 | -1.93 (0.22) | -2.36 (0.22)
  AM iTNSS Day 26: number analyzed (Participants) | 154 | 160
  AM iTNSS Day 26 | -2.10 (0.23) | -2.68 (0.22)
  AM iTNSS Day 27: number analyzed (Participants) | 144 | 152
  AM iTNSS Day 27 | -2.01 (0.23) | -2.49 (0.22)
  AM iTNSS Day 28: number analyzed (Participants) | 115 | 122
  AM iTNSS Day 28 | -1.96 (0.28) | -2.62 (0.26)
  rTNSS Day 1: number analyzed (Participants) | 167 | 176
  rTNSS Day 1 | -0.71 (0.16) | -0.93 (0.15)
  rTNSS Day 2: number analyzed (Participants) | 167 | 176
  rTNSS Day 2 | -0.91 (0.16) | -1.17 (0.16)
  rTNSS Day 3: number analyzed (Participants) | 167 | 176
  rTNSS Day 3 | -1.07 (0.17) | -1.38 (0.16)
  rTNSS Day 4: number analyzed (Participants) | 168 | 175
  rTNSS Day 4 | -1.15 (0.17) | -1.43 (0.16)
  rTNSS Day 5: number analyzed (Participants) | 168 | 176
  rTNSS Day 5 | -1.22 (0.17) | -1.35 (0.17)
  rTNSS Day 6: number analyzed (Participants) | 167 | 176
  rTNSS Day 6 | -1.21 (0.19) | -1.51 (0.18)
  rTNSS Day 7: number analyzed (Participants) | 168 | 174
  rTNSS Day 7 | -1.37 (0.19) | -1.66 (0.18)
  rTNSS Day 8: number analyzed (Participants) | 165 | 171
  rTNSS Day 8 | -1.58 (0.18) | -1.82 (0.18)
  rTNSS Day 9: number analyzed (Participants) | 165 | 171
  rTNSS Day 9 | -1.55 (0.20) | -1.92 (0.19)
  rTNSS Day 10: number analyzed (Participants) | 165 | 171
  rTNSS Day 10 | -1.60 (0.20) | -2.06 (0.19)
  rTNSS Day 11: number analyzed (Participants) | 162 | 169
  rTNSS Day 11 | -1.65 (0.20) | -1.96 (0.20)
  rTNSS Day 12: number analyzed (Participants) | 163 | 168
  rTNSS Day 12 | -1.81 (0.19) | -2.14 (0.19)
  rTNSS Day 13: number analyzed (Participants) | 162 | 168
  rTNSS Day 13 | -1.87 (0.20) | -2.12 (0.20)
  rTNSS Day 14: number analyzed (Participants) | 163 | 166
  rTNSS Day 14 | -1.83 (0.20) | -2.17 (0.20)
  rTNSS Day 15: number analyzed (Participants) | 163 | 165
  rTNSS Day 15 | -1.70 (0.20) | -2.11 (0.20)
  rTNSS Day 16: number analyzed (Participants) | 163 | 166
  rTNSS Day 16 | -1.82 (0.20) | -2.38 (0.20)
  rTNSS Day 17: number analyzed (Participants) | 163 | 166
  rTNSS Day 17 | -1.94 (0.21) | -2.53 (0.20)
  rTNSS Day 18: number analyzed (Participants) | 163 | 165
  rTNSS Day 18 | -2.21 (0.20) | -2.51 (0.20)
  rTNSS Day 19: number analyzed (Participants) | 162 | 166
  rTNSS Day 19 | -1.99 (0.20) | -2.44 (0.20)
  rTNSS Day 20: number analyzed (Participants) | 160 | 166
  rTNSS Day 20 | -2.16 (0.20) | -2.47 (0.20)
  rTNSS Day 21: number analyzed (Participants) | 159 | 166
  rTNSS Day 21 | -2.12 (0.21) | -2.54 (0.20)
  rTNSS Day 22: number analyzed (Participants) | 157 | 165
  rTNSS Day 22 | -2.01 (0.21) | -2.47 (0.21)
  rTNSS Day 23: number analyzed (Participants) | 159 | 165
  rTNSS Day 23 | -1.99 (0.21) | -2.30 (0.20)
  rTNSS Day 24: number analyzed (Participants) | 158 | 165
  rTNSS Day 24 | -2.12 (0.21) | -2.60 (0.20)
  rTNSS Day 25: number analyzed (Participants) | 158 | 164
  rTNSS Day 25 | -2.28 (0.22) | -2.44 (0.21)
  rTNSS Day 26: number analyzed (Participants) | 155 | 163
  rTNSS Day 26 | -2.25 (0.22) | -2.57 (0.21)
  rTNSS Day 27: number analyzed (Participants) | 149 | 154
  rTNSS Day 27 | -2.23 (0.22) | -2.51 (0.21)
  rTNSS Day 28: number analyzed (Participants) | 119 | 127
  rTNSS Day 28 | -1.93 (0.28) | -2.58 (0.26)
  AM rTNSS Day 1: number analyzed (Participants) | 165 | 174
  AM rTNSS Day 1 | -0.70 (0.18) | -1.02 (0.17)
  AM rTNSS Day 2: number analyzed (Participants) | 164 | 174
  AM rTNSS Day 2 | -0.97 (0.18) | -1.20 (0.17)
  AM rTNSS Day 3: number analyzed (Participants) | 167 | 176
  AM rTNSS Day 3 | -1.12 (0.18) | -1.37 (0.18)
  AM rTNSS Day 4: number analyzed (Participants) | 165 | 175
  AM rTNSS Day 4 | -1.11 (0.18) | -1.45 (0.18)
  AM rTNSS Day 5: number analyzed (Participants) | 165 | 174
  AM rTNSS Day 5 | -1.33 (0.19) | -1.48 (0.18)
  AM rTNSS Day 6: number analyzed (Participants) | 164 | 174
  AM rTNSS Day 6 | -1.30 (0.20) | -1.59 (0.20)
  AM rTNSS Day 7: number analyzed (Participants) | 157 | 168
  AM rTNSS Day 7 | -1.28 (0.21) | -1.69 (0.20)
  AM rTNSS Day 8: number analyzed (Participants) | 158 | 170
  AM rTNSS Day 8 | -1.74 (0.21) | -1.85 (0.20)
  AM rTNSS Day 9: number analyzed (Participants) | 160 | 171
  AM rTNSS Day 9 | -1.73 (0.21) | -1.94 (0.21)
  AM rTNSS Day 10: number analyzed (Participants) | 156 | 167
  AM rTNSS Day 10 | -1.65 (0.21) | -2.10 (0.20)
  AM rTNSS Day 11: number analyzed (Participants) | 160 | 166
  AM rTNSS Day 11 | -1.66 (0.21) | -1.96 (0.20)
  AM rTNSS Day 12: number analyzed (Participants) | 161 | 167
  AM rTNSS Day 12 | -1.82 (0.21) | -2.05 (0.20)
  AM rTNSS Day 13: number analyzed (Participants) | 156 | 163
  AM rTNSS Day 13 | -1.87 (0.22) | -2.06 (0.21)
  AM rTNSS Day 14: number analyzed (Participants) | 154 | 162
  AM rTNSS Day 14 | -1.84 (0.21) | -2.14 (0.20)
  AM rTNSS Day 15: number analyzed (Participants) | 156 | 163
  AM rTNSS Day 15 | -1.67 (0.22) | -2.15 (0.21)
  AM rTNSS Day 16: number analyzed (Participants) | 161 | 164
  AM rTNSS Day 16 | -1.75 (0.22) | -2.37 (0.21)
  AM rTNSS Day 17: number analyzed (Participants) | 161 | 160
  AM rTNSS Day 17 | -2.12 (0.22) | -2.62 (0.22)
  AM rTNSS Day 18: number analyzed (Participants) | 163 | 165
  AM rTNSS Day 18 | -2.22 (0.21) | -2.48 (0.21)
  AM rTNSS Day 19: number analyzed (Participants) | 159 | 164
  AM rTNSS Day 19 | -1.83 (0.22) | -2.37 (0.21)
  AM rTNSS Day 20: number analyzed (Participants) | 157 | 161
  AM rTNSS Day 20 | -2.18 (0.22) | -2.42 (0.22)
  AM rTNSS Day 21: number analyzed (Participants) | 152 | 163
  AM rTNSS Day 21 | -2.07 (0.22) | -2.64 (0.22)
  AM rTNSS Day 22: number analyzed (Participants) | 147 | 164
  AM rTNSS Day 22 | -2.02 (0.23) | -2.44 (0.22)
  AM rTNSS Day 23: number analyzed (Participants) | 158 | 162
  AM rTNSS Day 23 | -1.96 (0.23) | -2.17 (0.22)
  AM rTNSS Day 24: number analyzed (Participants) | 156 | 164
  AM rTNSS Day 24 | -2.03 (0.23) | -2.57 (0.22)
  AM rTNSS Day 25: number analyzed (Participants) | 158 | 163
  AM rTNSS Day 25 | -2.22 (0.23) | -2.45 (0.22)
  AM rTNSS Day 26: number analyzed (Participants) | 152 | 157
  AM rTNSS Day 26 | -2.19 (0.23) | -2.59 (0.23)
  AM rTNSS Day 27: number analyzed (Participants) | 145 | 153
  AM rTNSS Day 27 | -2.23 (0.23) | -2.54 (0.23)
  AM rTNSS Day 28: number analyzed (Participants) | 110 | 118
  AM rTNSS Day 28 | -1.82 (0.30) | -2.55 (0.27)
  PM rTNSS Day 1: number analyzed (Participants) | 144 | 152
  PM rTNSS Day 1 | -0.88 (0.20) | -0.97 (0.19)
  PM rTNSS Day 2: number analyzed (Participants) | 157 | 172
  PM rTNSS Day 2 | -0.91 (0.18) | -1.19 (0.17)
  PM rTNSS Day 3: number analyzed (Participants) | 159 | 170
  PM rTNSS Day 3 | -1.10 (0.19) | -1.39 (0.19)
  PM rTNSS Day 4: number analyzed (Participants) | 164 | 169
  PM rTNSS Day 4 | -1.17 (0.19) | -1.42 (0.19)
  PM rTNSS Day 5: number analyzed (Participants) | 164 | 172
  PM rTNSS Day 5 | -1.06 (0.19) | -1.29 (0.18)
  PM rTNSS Day 6: number analyzed (Participants) | 162 | 171
  PM rTNSS Day 6 | -1.13 (0.21) | -1.42 (0.20)
  PM rTNSS Day 7: number analyzed (Participants) | 164 | 168
  PM rTNSS Day 7 | -1.48 (0.20) | -1.64 (0.20)
  PM rTNSS Day 8: number analyzed (Participants) | 152 | 153
  PM rTNSS Day 8 | -1.34 (0.20) | -1.73 (0.19)
  PM rTNSS Day 9: number analyzed (Participants) | 158 | 166
  PM rTNSS Day 9 | -1.49 (0.21) | -1.89 (0.20)
  PM rTNSS Day 10: number analyzed (Participants) | 162 | 162
  PM rTNSS Day 10 | -1.58 (0.21) | -2.07 (0.21)
  PM rTNSS Day 11: number analyzed (Participants) | 157 | 162
  PM rTNSS Day 11 | -1.62 (0.22) | -2.02 (0.22)
  PM rTNSS Day 12: number analyzed (Participants) | 158 | 158
  PM rTNSS Day 12 | -1.86 (0.21) | -2.29 (0.21)
  PM rTNSS Day 13: number analyzed (Participants) | 151 | 166
  PM rTNSS Day 13 | -1.91 (0.22) | -2.18 (0.21)
  PM rTNSS Day 14: number analyzed (Participants) | 157 | 159
  PM rTNSS Day 14 | -1.85 (0.23) | -2.15 (0.22)
  PM rTNSS Day 15: number analyzed (Participants) | 146 | 155
  PM rTNSS Day 15 | -1.78 (0.22) | -2.15 (0.21)
  PM rTNSS Day 16: number analyzed (Participants) | 153 | 164
  PM rTNSS Day 16 | -1.84 (0.23) | -2.33 (0.22)
  PM rTNSS Day 17: number analyzed (Participants) | 159 | 158
  PM rTNSS Day 17 | -1.81 (0.22) | -2.51 (0.22)
  PM rTNSS Day 18: number analyzed (Participants) | 161 | 157
  PM rTNSS Day 18 | -2.22 (0.22) | -2.54 (0.23)
  PM rTNSS Day 19: number analyzed (Participants) | 156 | 162
  PM rTNSS Day 19 | -2.23 (0.21) | -2.53 (0.21)
  PM rTNSS Day 20: number analyzed (Participants) | 155 | 162
  PM rTNSS Day 20 | -2.17 (0.21) | -2.52 (0.20)
  PM rTNSS Day 21: number analyzed (Participants) | 152 | 160
  PM rTNSS Day 21 | -2.19 (0.23) | -2.48 (0.22)
  PM rTNSS Day 22: number analyzed (Participants) | 150 | 151
  PM rTNSS Day 22 | -2.03 (0.22) | -2.53 (0.22)
  PM rTNSS Day 23: number analyzed (Participants) | 150 | 161
  PM rTNSS Day 23 | -2.06 (0.23) | -2.41 (0.22)
  PM rTNSS Day 24: number analyzed (Participants) | 155 | 161
  PM rTNSS Day 24 | -2.25 (0.22) | -2.64 (0.21)
  PM rTNSS Day 25: number analyzed (Participants) | 153 | 161
  PM rTNSS Day 25 | -2.39 (0.23) | -2.42 (0.22)
  PM rTNSS Day 26: number analyzed (Participants) | 151 | 161
  PM rTNSS Day 26 | -2.31 (0.23) | -2.54 (0.22)
  PM rTNSS Day 27: number analyzed (Participants) | 147 | 149
  PM rTNSS Day 27 | -2.25 (0.23) | -2.54 (0.22)
  PM rTNSS Day 28: number analyzed (Participants) | 117 | 125
  PM rTNSS Day 28 | -2.07 (0.30) | -2.68 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 1; Test type: Superiority or Other; p = 0.011, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.450, 95% CI 2-sided [-0.80 to -0.10]
Statistical Analysis 2: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 2; Test type: Superiority or Other; p = 0.089, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.325, 95% CI 2-sided [-0.70 to 0.05]
Statistical Analysis 3: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 3; Test type: Superiority or Other; p = 0.052, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.393, 95% CI 2-sided [-0.79 to 0.00]
Statistical Analysis 4: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 4; Test type: Superiority or Other; p = 0.187, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.262, 95% CI 2-sided [-0.65 to 0.13]
Statistical Analysis 5: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 5; Test type: Superiority or Other; p = 0.164, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.298, 95% CI 2-sided [-0.72 to 0.12]
Statistical Analysis 6: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 6; Test type: Superiority or Other; p = 0.008, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.573, 95% CI 2-sided [-1.00 to -0.15]
Statistical Analysis 7: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 7; Test type: Superiority or Other; p = 0.082, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.376, 95% CI 2-sided [-0.80 to 0.05]
Statistical Analysis 8: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 8; Test type: Superiority or Other; p = 0.296, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.231, 95% CI 2-sided [-0.67 to 0.20]
Statistical Analysis 9: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 9; Test type: Superiority or Other; p = 0.383, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.191, 95% CI 2-sided [-0.62 to 0.24]
Statistical Analysis 10: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 10; Test type: Superiority or Other; p = 0.048, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.464, 95% CI 2-sided [-0.92 to -0.00]
Statistical Analysis 11: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 11; Test type: Superiority or Other; p = 0.469, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.172, 95% CI 2-sided [-0.64 to 0.29]
Statistical Analysis 12: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 12; Test type: Superiority or Other; p = 0.151, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.340, 95% CI 2-sided [-0.80 to 0.12]
Statistical Analysis 13: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 13; Test type: Superiority or Other; p = 0.145, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.344, 95% CI 2-sided [-0.81 to 0.12]
Statistical Analysis 14: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 14; Test type: Superiority or Other; p = 0.297, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.235, 95% CI 2-sided [-0.68 to 0.21]
Statistical Analysis 15: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 15; Test type: Superiority or Other; p = 0.094, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.380, 95% CI 2-sided [-0.82 to 0.07]
Statistical Analysis 16: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 16; Test type: Superiority or Other; p = 0.064, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.430, 95% CI 2-sided [-0.89 to 0.03]
Statistical Analysis 17: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 17; Test type: Superiority or Other; p = 0.019, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.563, 95% CI 2-sided [-1.03 to -0.09]
Statistical Analysis 18: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 18; Test type: Superiority or Other; p = 0.044, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.457, 95% CI 2-sided [-0.90 to -0.01]
Statistical Analysis 19: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 19; Test type: Superiority or Other; p = 0.007, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.633, 95% CI 2-sided [-1.09 to -0.17]
Statistical Analysis 20: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 20; Test type: Superiority or Other; p = 0.348, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.222, 95% CI 2-sided [-0.69 to 0.24]
Statistical Analysis 21: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 21; Test type: Superiority or Other; p = 0.243, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.281, 95% CI 2-sided [-0.76 to 0.19]
Statistical Analysis 22: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 22; Test type: Superiority or Other; p = 0.014, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.595, 95% CI 2-sided [-1.07 to -0.12]
Statistical Analysis 23: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 23; Test type: Superiority or Other; p = 0.055, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.474, 95% CI 2-sided [-0.96 to 0.01]
Statistical Analysis 24: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 24; Test type: Superiority or Other; p = 0.062, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.464, 95% CI 2-sided [-0.95 to 0.02]
Statistical Analysis 25: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 25; Test type: Superiority or Other; p = 0.079, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.430, 95% CI 2-sided [-0.91 to 0.05]
Statistical Analysis 26: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 26; Test type: Superiority or Other; p = 0.019, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.576, 95% CI 2-sided [-1.06 to -0.10]
Statistical Analysis 27: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 27; Test type: Superiority or Other; p = 0.056, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.480, 95% CI 2-sided [-0.97 to 0.01]
Statistical Analysis 28: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM iTNSS at Day 28; Test type: Superiority or Other; p = 0.018, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.659, 95% CI 2-sided [-1.20 to -0.11]
Statistical Analysis 29: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 1; Test type: Superiority or Other; p = 0.194, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.222, 95% CI 2-sided [-0.56 to 0.1]
Statistical Analysis 30: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 2; Test type: Superiority or Other; p = 0.134, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.263, 95% CI 2-sided [-0.61 to 0.08]
Statistical Analysis 31: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 3; Test type: Superiority or Other; p = 0.091, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.310, 95% CI 2-sided [-0.67 to 0.05]
Statistical Analysis 32: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 4; Test type: Superiority or Other; p = 0.131, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.278, 95% CI 2-sided [-0.64 to 0.08]
Statistical Analysis 33: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 5; Test type: Superiority or Other; p = 0.483, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.130, 95% CI 2-sided [-0.49 to 0.23]
Statistical Analysis 34: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 6; Test type: Superiority or Other; p = 0.137, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.301, 95% CI 2-sided [-0.70 to 0.10]
Statistical Analysis 35: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 7; Test type: Superiority or Other; p = 0.142, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.297, 95% CI 2-sided [-0.69 to 0.10]
Statistical Analysis 36: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 8; Test type: Superiority or Other; p = 0.220, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.245, 95% CI 2-sided [-0.64 to 0.15]
Statistical Analysis 37: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 9; Test type: Superiority or Other; p = 0.081, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.373, 95% CI 2-sided [-0.79 to 0.05]
Statistical Analysis 38: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 10; Test type: Superiority or Other; p = 0.034, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.453, 95% CI 2-sided [-0.87 to -0.04]
Statistical Analysis 39: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 11; Test type: Superiority or Other; p = 0.150, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.314, 95% CI 2-sided [-0.74 to 0.11]
Statistical Analysis 40: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 12; Test type: Superiority or Other; p = 0.111, ANCOVA; Mean Difference (Net) = -0.333, 95% CI 2-sided [-0.74 to 0.08]
Statistical Analysis 41: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 13; Test type: Superiority or Other; p = 0.261, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.250, 95% CI 2-sided [-0.69 to 0.19]
Statistical Analysis 42: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 14; Test type: Superiority or Other; p = 0.123, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.342, 95% CI 2-sided [-0.78 to 0.09]
Statistical Analysis 43: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 15; Test type: Superiority or Other; p = 0.056, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.415, 95% CI 2-sided [-0.84 to 0.01]
Statistical Analysis 44: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 16; Test type: Superiority or Other; p = 0.011, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.566, 95% CI 2-sided [-1.00 to -0.13]
Statistical Analysis 45: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 17; Test type: Superiority or Other; p = 0.009, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.590, 95% CI 2-sided [-1.03 to -0.15]
Statistical Analysis 46: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 18; Test type: Superiority or Other; p = 0.175, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.301, 95% CI 2-sided [-0.74 to 0.13]
Statistical Analysis 47: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 19; Test type: Superiority or Other; p = 0.039, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.449, 95% CI 2-sided [-0.87 to -0.02]
Statistical Analysis 48: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 20; Test type: Superiority or Other; p = 0.152, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.315, 95% CI 2-sided [-0.75 to 0.12]
Statistical Analysis 49: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 21; Test type: Superiority or Other; p = 0.063, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.424, 95% CI 2-sided [-0.87 to 0.02]
Statistical Analysis 50: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 22; Test type: Superiority or Other; p = 0.044, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.454, 95% CI 2-sided [-0.90 to -0.01]
Statistical Analysis 51: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 23; Test type: Superiority or Other; p = 0.179, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.312, 95% CI 2-sided [-0.77 to 0.14]
Statistical Analysis 52: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 24; Test type: Superiority or Other; p = 0.034, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.479, 95% CI 2-sided [-0.92 to -0.04]
Statistical Analysis 53: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 25; Test type: Superiority or Other; p = 0.505, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.157, 95% CI 2-sided [-0.62 to 0.31]
Statistical Analysis 54: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 26; Test type: Superiority or Other; p = 0.186, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.317, 95% CI 2-sided [-0.79 to 0.15]
Statistical Analysis 55: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 27; Test type: Superiority or Other; p = 0.234, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.283, 95% CI 2-sided [-0.75 to 0.18]
Statistical Analysis 56: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for rTNSS at Day 28; Test type: Superiority or Other; p = 0.017, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.645, 95% CI 2-sided [-1.17 to -0.12]
Statistical Analysis 57: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 1; Test type: Superiority or Other; p = 0.095, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.320, 95% CI 2-sided [-0.70 to 0.06]
Statistical Analysis 58: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 2; Test type: Superiority or Other; p = 0.236, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.231, 95% CI 2-sided [-0.61 to 0.15]
Statistical Analysis 59: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 3; Test type: Superiority or Other; p = 0.205, ANCOVA; Mean Difference (Net) = -0.255, 95% CI 2-sided [-0.65 to 0.14]
Statistical Analysis 60: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 4; Test type: Superiority or Other; p = 0.084, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.343, 95% CI 2-sided [-0.73 to 0.05]
Statistical Analysis 61: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 5; Test type: Superiority or Other; p = 0.475, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.146, 95% CI 2-sided [-0.55 to 0.26]
Statistical Analysis 62: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 6; Test type: Superiority or Other; p = 0.178, ANCOVA; Mean Difference (Net) = -0.296, 95% CI 2-sided [-0.73 to 0.14]
Statistical Analysis 63: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 7; Test type: Superiority or Other; p = 0.071, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.406, 95% CI 2-sided [-0.85 to 0.04]
Statistical Analysis 64: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 8; Test type: Superiority or Other; p = 0.621, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.111, 95% CI 2-sided [-0.55 to 0.33]
Statistical Analysis 65: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 9; Test type: Superiority or Other; p = 0.372, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.206, 95% CI 2-sided [-0.66 to 0.25]
Statistical Analysis 66: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 10; Test type: Superiority or Other; p = 0.046, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.452, 95% CI 2-sided [-0.90 to -0.01]
Statistical Analysis 67: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 11; Test type: Superiority or Other; p = 0.183, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.302, 95% CI 2-sided [-0.75 to 0.14]
Statistical Analysis 68: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 12; Test type: Superiority or Other; p = 0.320, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.226, 95% CI 2-sided [-0.67 to 0.22]
Statistical Analysis 69: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 13; Test type: Superiority or Other; p = 0.431, ANCOVA; Mean Difference (Net) = -0.188, 95% CI 2-sided [-0.66 to 0.28]
Statistical Analysis 70: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 14; Test type: Superiority or Other; p = 0.191, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.299, 95% CI 2-sided [-0.75 to 0.15]
Statistical Analysis 71: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 15; Test type: Superiority or Other; p = 0.043, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.475, 95% CI 2-sided [-0.94 to -0.02]
Statistical Analysis 72: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 16; Test type: Superiority or Other; p = 0.009, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.619, 95% CI 2-sided [-1.08 to -0.16]
Statistical Analysis 73: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 17; Test type: Superiority or Other; p = 0.040, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.495, 95% CI 2-sided [-0.97 to -0.02]
Statistical Analysis 74: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 18; Test type: Superiority or Other; p = 0.249, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.262, 95% CI 2-sided [-0.71 to 0.18]
Statistical Analysis 75: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 19; Test type: Superiority or Other; p = 0.023, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.536, 95% CI 2-sided [-1.00 to -0.07]
Statistical Analysis 76: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 20; Test type: Superiority or Other; p = 0.321, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.240, 95% CI 2-sided [-0.71 to 0.23]
Statistical Analysis 77: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 21; Test type: Superiority or Other; p = 0.019, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.568, 95% CI 2-sided [-1.04 to -0.09]
Statistical Analysis 78: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 22; Test type: Superiority or Other; p = 0.092, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.419, 95% CI 2-sided [-0.91 to 0.07]
Statistical Analysis 79: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 23; Test type: Superiority or Other; p = 0.404, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.206, 95% CI 2-sided [-0.69 to 0.28]
Statistical Analysis 80: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 24; Test type: Superiority or Other; p = 0.027, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.546, 95% CI 2-sided [-1.03 to -0.06]
Statistical Analysis 81: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 25; Test type: Superiority or Other; p = 0.357, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.227, 95% CI 2-sided [-0.71 to 0.26]
Statistical Analysis 82: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 26; Test type: Superiority or Other; p = 0.114, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.403, 95% CI 2-sided [-0.90 to 0.10]
Statistical Analysis 83: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 27; Test type: Superiority or Other; p = 0.228, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.307, 95% CI 2-sided [-0.81 to 0.19]
Statistical Analysis 84: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for AM rTNSS at Day 28; Test type: Superiority or Other; p = 0.012, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.725, 95% CI 2-sided [-1.29 to -0.16]
Statistical Analysis 85: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 1; Test type: Superiority or Other; p = 0.643, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.093, 95% CI 2-sided [-0.49 to 0.30]
Statistical Analysis 86: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 2; Test type: Superiority or Other; p = 0.150, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.279, 95% CI 2-sided [-0.66 to 0.10]
Statistical Analysis 87: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 3; Test type: Superiority or Other; p = 0.162, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.291, 95% CI 2-sided [-0.70 to 0.12]
Statistical Analysis 88: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 4; Test type: Superiority or Other; p = 0.242, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.244, 95% CI 2-sided [-0.65 to 0.17]
Statistical Analysis 89: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 5; Test type: Superiority or Other; p = 0.278, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.223, 95% CI 2-sided [-0.63 to 0.18]
Statistical Analysis 90: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 6; Test type: Superiority or Other; p = 0.200, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.282, 95% CI 2-sided [-0.71 to 0.15]
Statistical Analysis 91: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 7; Test type: Superiority or Other; p = 0.456, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.164, 95% CI 2-sided [-0.60 to 0.27]
Statistical Analysis 92: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 8; Test type: Superiority or Other; p = 0.076, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.385, 95% CI 2-sided [-0.81 to 0.04]
Statistical Analysis 93: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 9; Test type: Superiority or Other; p = 0.084, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.396, 95% CI 2-sided [-0.85 to 0.05]
Statistical Analysis 94: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 10; Test type: Superiority or Other; p = 0.040, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.481, 95% CI 2-sided [-0.94 to -0.02]
Statistical Analysis 95: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 11; Test type: Superiority or Other; p = 0.090, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.405, 95% CI 2-sided [-0.87 to 0.06]
Statistical Analysis 96: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 12; Test type: Superiority or Other; p = 0.060, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.432, 95% CI 2-sided [-0.88 to 0.02]
Statistical Analysis 97: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 13; Test type: Superiority or Other; p = 0.252, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.277, 95% CI 2-sided [-0.75 to 0.20]
Statistical Analysis 98: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 14; Test type: Superiority or Other; p = 0.229, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.300, 95% CI 2-sided [-0.79 to 0.19]
Statistical Analysis 99: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 15; Test type: Superiority or Other; p = 0.109, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.373, 95% CI 2-sided [-0.83 to 0.08]
Statistical Analysis 100: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 16; Test type: Superiority or Other; ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.484, 95% CI 2-sided [-0.96 to -0.01]
Statistical Analysis 101: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 17; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.700, 95% CI 2-sided [-1.17 to -0.23]
Statistical Analysis 102: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 18; Test type: Superiority or Other; p = 0.182, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.326, 95% CI 2-sided [-0.81 to 0.15]
Statistical Analysis 103: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 19; Test type: Superiority or Other; p = 0.194, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.299, 95% CI 2-sided [-0.75 to 0.15]
Statistical Analysis 104: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 20; Test type: Superiority or Other; p = 0.129, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.348, 95% CI 2-sided [-0.80 to 0.10]
Statistical Analysis 105: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 21; Test type: Superiority or Other; p = 0.232, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.292, 95% CI 2-sided [-0.77 to 0.19]
Statistical Analysis 106: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 22; Test type: Superiority or Other; p = 0.042, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.499, 95% CI 2-sided [-0.98 to -0.02]
Statistical Analysis 107: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 23; Test type: Superiority or Other; p = 0.150, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.356, 95% CI 2-sided [-0.84 to 0.13]
Statistical Analysis 108: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 24; Test type: Superiority or Other; p = 0.090, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.398, 95% CI 2-sided [-0.86 to 0.06]
Statistical Analysis 109: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 25; Test type: Superiority or Other; p = 0.909, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.028, 95% CI 2-sided [-0.52 to 0.46]
Statistical Analysis 110: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 26; Test type: Superiority or Other; p = 0.354, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.233, 95% CI 2-sided [-0.73 to 0.26]
Statistical Analysis 111: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 27; Test type: Superiority or Other; p = 0.245, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.290, 95% CI 2-sided [-0.78 to 0.20]
Statistical Analysis 112: Comparison: Placebo vs Fluticasone Furoate 110 mcg QD; Placebo versus Fluticasone Furoate 110 mcg QD for PM rTNSS at Day 28; Test type: Superiority or Other; p = 0.038, ANCOVA; ANCOVA method was used adjusting for baseline rTNSS, country, age, and gender, in addition to treatment effect; Mean Difference (Net) = -0.601, 95% CI 2-sided [-1.17 to -0.03]

ADVERSE EVENTS:
Time Frame: AEs were collected from screening up to 32 days
Description: ITT Population (participants who were randomized and received at least one dose of study drug was used for the analysis of serious adverse event (SAE) and non-serious AEs. Non-serious AEs have been reported for the treatment period (28 days).
Arm/Group | Placebo | Fluticasone Furoate 110mcg QD
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/179
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/179
Other Adverse Events (participants affected / at risk) | 65/173 | 61/179
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=173) | Fluticasone Furoate 110mcg QD (N=179)
Headache (Nervous system disorders) | 23 | 12
Sinus headache (Nervous system disorders) | 3 | 2
Migraine (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 1 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Perianal abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dry eye (Eye disorders) | 2 | 2
Conjunctivitis (Eye disorders) | 2 | 0
Eye pruritus (Eye disorders) | 0 | 2
Conjunctival oedema (Eye disorders) | 1 | 0
Lacrimation decreased (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1
Blood pressure increased (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.